CLINICAL TRIAL: NCT04356859
Title: The Acute Burn ResUscitation Multicenter Prospective Trial (ABRUPT2)
Brief Title: The Acute Burn ResUscitation Multicenter Prospective Trial
Acronym: ABRUPT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Burn Association (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1528946; CDMRP-JW180038 (Other Grant/Funding Number: US Army Department of Defense CDMRP)
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Burn Injury
Keywords: Resuscitation
MeSH Terms: conditions — Burns | interventions — Serum Albumin, Human; Albumins

STUDY DESIGN:
Intervention Model Description: Randomization will be based on "intent to treat." Consecutively admitted and eligible burn patients will be assigned to one of two treatment groups (Colloid or Crystalloid) within 12 hours of burn injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid (No Intervention): Subjects in the crystalloid group will receive fluid resuscitation with Lactated Ringer's titrated each hour to achieve a urine output of 0.5-1mL/kg predicted body weight.
- Colloid (Active Comparator): Subjects in the colloid group will receive fluid resuscitation with Lactated Ringer's and 5% human albumin solution introduced no earlier than 8 hours post burn and no later than 12 hours post burn in a ratio by volume of 1/3 albumin to 2/3 Lactated Ringer's, and titrated each hour to achieve a urine output of 0.5-1mL/kg (milliliter/kilogram) predicted body weight.
  Interventions: Drug: Albumin Human

INTERVENTIONS:
Drug: Albumin Human — Addition of albumin during acute resuscitation following burn injury
  Other Names: albumin
  Arms: Colloid

SUMMARY:
This is a prospective randomized multi-center study which will compare acute fluid resuscitation using a colloid strategy (LR + 5% Albumin) to a crystalloid strategy (LR alone), in adults with an acute burn involving at least 25% of their total body surface area.

DETAILED DESCRIPTION:
Enrolled subjects will be randomly assigned to either the Colloid Group or the Crystalloid Group. Randomization will be based on an intent-to-treat basis. In order to ensure that the two groups have comparable injury severity at baseline, randomization will be block- stratified based on age (18-50 and > 50 years), burn size (25-50% and > 50% TBSA), and presence of inhalation injury confirmed by bronchoscopy (present or absent). In the Colloid Group resuscitation starts with LR and then 5% albumin will be introduced between 8 and 12 hours post burn in a ratio of 1/3 albumin to 2/3 LR. In the Crystalloid Group resuscitation is with LR only. Each group will have their study fluid maintained for the 1st 48 hours post burn and study fluids in each group will be identically titrated to the urinary output.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Total burn size (second and third degree) is ≥ 25% of the TBSA
* Burn center admission within 12 hours of injury.
* There is a plan for formal fluid resuscitation.

Exclusion Criteria:

* Significant associated trauma
* High voltage (≥ 1000 volts) electrical burns
* Burn wound excision surgery within 48 hours from injury
* Fresh frozen plasma (FFP) given at any time ≤ 48 hours from injury
* Hypertonic saline (HTS) given at any time ≤ 48 hours from injury
* Hydroxyethyl starch (HES) given at any time ≤ 48 hours from injury
* High dose Vitamin C infusion given at any time ≤ 48 hours from injury
* Administration of human albumin prior to randomization
* Palliative comfort measures are instituted ≤ 48 hours from injury
* Pregnancy
* Pre-injury chronic renal insufficiency equal to or greater than stage 3
* Pre-injury chronic hepatic disease (Child-Pugh B or C)
* Pre-injury left ventricular (LV) dysfunction (echocardiography LV grade II-IV or ejection fraction ≤ 35%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Volume of fluid received during resuscitation for burn injury | 24 hours post burn injury
  Total fluid resuscitation volume at 24 hours post burn in mL/kg/% TBSA burn

SECONDARY OUTCOMES:
Volume of fluid received during resuscitation for burn injury | 48 hours post burn injury
  Total resuscitation volume at 48 hours in mL/kg/%TBSA burn.
Urine output during resuscitation for burn injury | 24 and 48 hours post burn injury
  Mean hourly urine output during resuscitation for burn injury
Number of crossovers | 48 hours post burn injury
  Number of crossovers between study arms during resuscitation for burn injury
Peak lactate and delta lactate | 48 hours post burn injury
  peak lactate level and delta lactate (peak lactate minus admission lactate)
Peak intra-abdominal pressure (IAP) and delta IAP | 48 hours post burn injury
  Peak intra-abdominal pressure (IAP) and delta IAP (peak IAP minus admission IAP)
Occurrence of Abdominal compartment syndrome | 48 hours post burn injury
  Abdominal compartment syndrome during resuscitation for burn injury
Occurrence of Limb or abdominal fasciotomy | 48 hours post burn injury
  Limb or abdominal fasciotomy during resuscitation for burn injury
Sequential Organ Failure Assessment (SOFA) score | 48, 72, and 96 hours post burn injury
  Assessment of organ function or failure by Sequential Organ Failure Assessment (SOFA)score, with the higher score(s) indicating organ failure
Acute kidney injury (AKI) | 96 hours post burn injury
  Diagnosis of AKI
Duration of intubation/mechanical ventilation | 96 hours post burn injury
  Duration of intubation/mechanical ventilation
PaO2/FiO2 ratios | 24, 48, 72, and 96 hours post burn injury
  PaO2(partial pressure of oxygen)/FiO2(fraction of inspired oxygen inspired oxygen) ratios
Time to wound healing | 7 days post last surgery for grafting of burn injury
  Time to wound healing defined as 7 days post last grafting surgery
Survival | 28 days post injury and hospital discharge
  28 day survival and hospital stay survival

CONTACTS AND LOCATIONS:
Overall Officials: David G Greenhalgh, MD, Principal Investigator — UC Davis Health
Locations (26):
- United States (24):
  - Arizona Burn Center Valleywise Health, Phoenix, Arizona
  - University of California Davis, Regional Burn Center, Sacramento, California
  - Torrance Memorial, Torrance, California
  - University of Florida Health, Gainesville, Florida
  - University of Miami Health System, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Loyola Medicine, Maywood, Illinois
  - University of Iowa Healthcare, Iowa City, Iowa
  - University of Kansas Health System, Kansas City, Kansas
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Westchester Medical Center Health Network, Valhalla, New York
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Legacy Health, Portland, Oregon
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Utah Health, Salt Lake City, Utah
  - Regional Burn Center at Harborview, Seattle, Washington
  - University of Wisconsin Health, Madison, Wisconsin
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pruitt BA Jr. Protection from excessive resuscitation: "pushing the pendulum back". J Trauma. 2000 Sep;49(3):567-8. doi: 10.1097/00005373-200009000-00030. No abstract available. PMID 11003341
- [Background] Zak AL, Harrington DT, Barillo DJ, Lawlor DF, Shirani KZ, Goodwin CW. Acute respiratory failure that complicates the resuscitation of pediatric patients with scald injuries. J Burn Care Rehabil. 1999 Sep-Oct;20(5):391-9. doi: 10.1097/00004630-199909000-00011. PMID 10501327
- [Background] Hobson KG, Young KM, Ciraulo A, Palmieri TL, Greenhalgh DG. Release of abdominal compartment syndrome improves survival in patients with burn injury. J Trauma. 2002 Dec;53(6):1129-33; discussion 1133-4. doi: 10.1097/00005373-200212000-00016. PMID 12478039
- [Background] Klein MB, Hayden D, Elson C, Nathens AB, Gamelli RL, Gibran NS, Herndon DN, Arnoldo B, Silver G, Schoenfeld D, Tompkins RG. The association between fluid administration and outcome following major burn: a multicenter study. Ann Surg. 2007 Apr;245(4):622-8. doi: 10.1097/01.sla.0000252572.50684.49. PMID 17414612
- [Background] Recinos PR, Hartford CA, Ziffren SE. Fluid resuscitation of burn patients comparing a crystalloid with a colloid containing solution: a prospective study. J Iowa Med Soc. 1975 Oct;65(10):426-32. No abstract available. PMID 1194720
- [Background] Goodwin CW, Dorethy J, Lam V, Pruitt BA Jr. Randomized trial of efficacy of crystalloid and colloid resuscitation on hemodynamic response and lung water following thermal injury. Ann Surg. 1983 May;197(5):520-31. doi: 10.1097/00000658-198305000-00004. PMID 6342554
- [Background] Cooper AB, Cohn SM, Zhang HS, Hanna K, Stewart TE, Slutsky AS; ALBUR Investigators. Five percent albumin for adult burn shock resuscitation: lack of effect on daily multiple organ dysfunction score. Transfusion. 2006 Jan;46(1):80-9. doi: 10.1111/j.1537-2995.2005.00667.x. PMID 16398734
- [Background] O'Mara MS, Slater H, Goldfarb IW, Caushaj PF. A prospective, randomized evaluation of intra-abdominal pressures with crystalloid and colloid resuscitation in burn patients. J Trauma. 2005 May;58(5):1011-8. doi: 10.1097/01.ta.0000162732.39083.15. PMID 15920417
- [Background] Muller Dittrich MH, Brunow de Carvalho W, Lopes Lavado E. Evaluation of the "Early" Use of Albumin in Children with Extensive Burns: A Randomized Controlled Trial. Pediatr Crit Care Med. 2016 Jun;17(6):e280-6. doi: 10.1097/PCC.0000000000000728. PMID 27077832
- [Background] Cartotto R, Callum J. A review of the use of human albumin in burn patients. J Burn Care Res. 2012 Nov-Dec;33(6):702-17. doi: 10.1097/BCR.0b013e31825b1cf6. PMID 23143614
- [Background] Baxter CR, Shires T. Physiological response to crystalloid resuscitation of severe burns. Ann N Y Acad Sci. 1968 Aug 14;150(3):874-94. doi: 10.1111/j.1749-6632.1968.tb14738.x. No abstract available. PMID 4973463
- [Background] Pruitt BA Jr. Fluid and electrolyte replacement in the burned patient. Surg Clin North Am. 1978 Dec;58(6):1291-1312. doi: 10.1016/s0039-6109(16)41692-0. No abstract available. PMID 734610
- [Background] Pruitt BA Jr. The burn patient: II. Later care and complications of thermal injury. Curr Probl Surg. 1979 May;16(5):1-95. doi: 10.1016/s0011-3840(79)80009-x. PMID 376227
- [Background] Cartotto RC, Innes M, Musgrave MA, Gomez M, Cooper AB. How well does the Parkland formula estimate actual fluid resuscitation volumes? J Burn Care Rehabil. 2002 Jul-Aug;23(4):258-65. doi: 10.1097/00004630-200207000-00006. PMID 12142578
- [Background] Cartotto R, Zhou A. Fluid creep: the pendulum hasn't swung back yet! J Burn Care Res. 2010 Jul-Aug;31(4):551-8. doi: 10.1097/BCR.0b013e3181e4d732. PMID 20616649
- [Background] Engrav LH, Colescott PL, Kemalyan N, Heimbach DM, Gibran NS, Solem LD, Dimick AR, Gamelli RL, Lentz CW. A biopsy of the use of the Baxter formula to resuscitate burns or do we do it like Charlie did it? J Burn Care Rehabil. 2000 Mar-Apr;21(2):91-5. doi: 10.1097/00004630-200021020-00002. PMID 10752739
- [Background] Cancio LC, Chavez S, Alvarado-Ortega M, Barillo DJ, Walker SC, McManus AT, Goodwin CW. Predicting increased fluid requirements during the resuscitation of thermally injured patients. J Trauma. 2004 Feb;56(2):404-13; discussion 413-4. doi: 10.1097/01.TA.0000075341.43956.E4. PMID 14960986
- [Background] Saffle JI. The phenomenon of "fluid creep" in acute burn resuscitation. J Burn Care Res. 2007 May-Jun;28(3):382-95. doi: 10.1097/BCR.0B013E318053D3A1. PMID 17438489
- [Background] Jelenko C 3rd, Williams JB, Wheeler ML, Callaway BD, Fackler VK, Albers CA, Barger AA. Studies in shock and resuscitation, I: use of a hypertonic, albumin-containing, fluid demand regimen (HALFD) in resuscitation. Crit Care Med. 1979 Apr;7(4):157-67. PMID 446052
- [Background] Lawrence A, Faraklas I, Watkins H, Allen A, Cochran A, Morris S, Saffle J. Colloid administration normalizes resuscitation ratio and ameliorates "fluid creep". J Burn Care Res. 2010 Jan-Feb;31(1):40-7. doi: 10.1097/BCR.0b013e3181cb8c72. PMID 20061836
- [Background] Faraklas I, Lam U, Cochran A, Stoddard G, Saffle J. Colloid normalizes resuscitation ratio in pediatric burns. J Burn Care Res. 2011 Jan-Feb;32(1):91-7. doi: 10.1097/BCR.0b013e318204b379. PMID 21131844
- [Background] Mehrkens HH, Ahnefeld FW. Volume and fluid replacement in the early post burn period: an animal experimental study. Burns 1979;5:113-15
- [Background] Asch MJ, Feldman RJ, Walker HL, Foley FD, Popp RL, Mason AD Jr, Pruitt BA Jr. Systemic and pulmonary hemodynamic changes accompanying thermal injury. Ann Surg. 1973 Aug;178(2):218-21. doi: 10.1097/00000658-197308000-00020. No abstract available. PMID 4723430
- [Background] Demling RH, Kramer G, Harms B. Role of thermal injury-induced hypoproteinemia on fluid flux and protein permeability in burned and nonburned tissue. Surgery. 1984 Feb;95(2):136-44. PMID 6695330
- [Background] Demling RH, Kramer GC, Gunther R, Nerlich M. Effect of nonprotein colloid on postburn edema formation in soft tissues and lung. Surgery. 1984 May;95(5):593-602. PMID 6200946
- [Background] Onarheim H, Reed RK. Thermal skin injury: effect of fluid therapy on the transcapillary colloid osmotic gradient. J Surg Res. 1991 Mar;50(3):272-8. doi: 10.1016/0022-4804(91)90190-w. PMID 1999916
- [Background] Moncrief JA. Effect of various fluid regimens and pharmacologic agents on the circulatory hemodynamics of the immediate postburn period. Ann Surg. 1966 Oct;164(4):723-52. doi: 10.1097/00000658-196610000-00017. No abstract available. PMID 5924792
- [Background] Park SH, Hemmila MR, Wahl WL. Early albumin use improves mortality in difficult to resuscitate burn patients. J Trauma Acute Care Surg. 2012 Nov;73(5):1294-7. doi: 10.1097/TA.0b013e31827019b1. PMID 23117385